CLINICAL TRIAL: NCT01907698
Title: Effect of Vaginal Intercourse on Spontaneous Labour at Term- A Randomized Trial
Brief Title: Effect of Vaginal Intercourse on Spontaneous Labour at Term
Status: Completed | Type: Observational
Sponsor: Hospital de Santa Maria, Portugal (Other)
Responsible Party: Principal Investigator, Catarina Castro, Dr, Hospital de Santa Maria, Portugal
Other Study IDs: Catarina Castro
Record Dates: First submitted 2013-07-05; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Spontaneous Labour Onset; Vaginal Intercourse at Term
Keywords: vaginal intercourse; labour; term pregnancy
MeSH Terms: conditions — Coitus | interventions — Sex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Vaginal coitus group: Pregnant women assigned to have vaginal coitus at least twice a week
  Interventions: Behavioral: Vaginal intercourse
- Control group: Pregnant women assigned to have no vaginal intercourse

INTERVENTIONS:
Behavioral: Vaginal intercourse — vaginal intercourse at least twice a week
  Groups: Vaginal coitus group

SUMMARY:
Vaginal intercourse to promote labour onset is biologically plausible. Oxytocin release during female orgasm, cervix mechanical stimulation and the effect of semen's prostaglandins are possible involved mechanisms. The investigators propose to evaluate the effect of vaginal intercourse on spontaneous labour at term.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnancy
* Singleton pregnancy
* Cephalic presentation
* No previous cesarean section
* Irrelevant obstetric history
* Surveiled pregnancy without complications

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pregnant women attending to antenatal appointment in our Obstetric Unit
Sampling Method: Probability Sample
Enrollment: 123 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Spontaneous labour onset at term | Spontaneous labour onset between 37 and 42 weeks of pregnancy
  Spontaneous labour was considered to be established when there were regular contractions and at least 3cm of cervical dilation.

SECONDARY OUTCOMES:
Gestational age at delivery | Gestational age at delivery (between 37 and 42 weeks of pregnancy)
Mode of delivery | Mode of delivery (vaginal or cesarean delivery) up to 42 weeks of pregnancy
  Route of delivery - vaginally or cesarean
Interval between recruitment and delivery | number of days between patients study recruitment and delivery (maximum period of 28 days - between 38 and 41/0-6 weeks/days of pregnancy)
  number of days between patients study recruitment and delivery (patients were included in the study at 38 weeks of pregnancy and followed until delivery; if spontaneous labour did not occur labour induction was scheduled during the 41th week of pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Catarina Castro, Dr, Principal Investigator — Hospital de Santa Maria
Locations (1):
- Hospital de Santa Maria, Lisbon, Portugal

REFERENCES:
- [Derived] Castro C, Afonso M, Carvalho R, Clode N, Graca LM. Effect of vaginal intercourse on spontaneous labor at term: a randomized controlled trial. Arch Gynecol Obstet. 2014 Dec;290(6):1121-5. doi: 10.1007/s00404-014-3343-0. Epub 2014 Jul 18. PMID 25033717